CLINICAL TRIAL: NCT03243019
Title: Evaluation of the Efficacy of Rapamycin in the Treatment of Cervico-facial Lymphatic Malformations of Poor Prognosis
Brief Title: Efficacy of Rapamycin in the Treatment of Cervico-facial Lymphatic Malformations
Acronym: RAPAMALYMPH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012_67; 2013-002800-15 (EudraCT Number)
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lymphatic Malformation; Pediatric
Keywords: cervico-facial; rapamycin
MeSH Terms: conditions — Lymphatic Abnormalities | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIROLIMUS (Experimental)
  Interventions: Drug: rapamycin; Device: MRI; Biological: Rapamycin dosage

INTERVENTIONS:
Drug: rapamycin — oral administration
Device: MRI — cervicofacial MRI
Biological: Rapamycin dosage — Biological dosage of Rapamycin level

SUMMARY:
To evaluate the efficacy of Rapamycin in extended cervicofacial lymphatic malformations in pediatric patients. Rapamycin is administered oral for a 6 month period.

The success rate is determined by volume reduction superior to 1/5e of the initial volume measured by MRI, impact on QOL and reduction of bleeding in case of mucosal involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 0 to 18 years of age, presenting with poly-cystic suprahyoid or mediastinal lymphatic.
* with chronic pain or functional respiratory or swallowing impairment with a CDS score < 8
* Curative treatment is not possible or associated with a high risk of morbidity ,mortality and functional and cosmetic impairment
* Karnofsky Score (> 10 years of age) or Lansky score (≤10 years of age) > 50%
* Biology

  * Neutrophils count≥1.0 x 109/L
  * Platelets count ≥ 100 x 109/L
  * Hemoglobin ≥ 8 g/dL
  * Bilirubin ≤ 1,5 ULN
  * Transaminases < 2,5 ULN
  * Serum albumin ≥ 2 g/dL.
  * LDL cholesterol <160 mg/dL
  * Triglycerides < 150 mg/dL
* Negative test of pregnancy if relevant
* Social security affiliation
* At least 2 months after a previous procedure on the malformation

Exclusion Criteria:

* Non-respect of inclusion criteria
* Other immunosuppressive therapy or long-term general corticosteroid therapy without a 28-day washout period
* renal failure
* Liver failure
* Digestive disease leading to rapamycin malabsorption
* uncontrolled or severe infectious disease
* Patients requiring treatment interfering with CYP3A4 isoenzyme (rifampicin, rifabutin, carbamazepine, phenobarbital, phenytoin) or inhibiting CYP3A4 isoenzyme's activity (ketoconazole, voriconazole, itraconazole, telithromycin, clarithromycin, Diltiazem, Verapamil, nicardipine, clotrimazole, fluconazole , troleandomycin, bromocriptine, cimetidine, danazol, protease inhibitors) -patients requiring treatment by cisapride and metoclopramide
* Concomitant administration of mTOR inhibitor
* Peanuts or soya allergy
* Impossibility to receive informed consent
* Absence of social security affiliation
* refusal to sign consent
* Ongoing pregnancy or breastfeeding
* refusal to participate

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Response rate to rapamycin | At 3 months
  Volumetric assessment by MRI. A response is considered as positive if volume decrease is superior to 1/5th of the initial volume.

SECONDARY OUTCOMES:
Kinetic of rapamycin response | At 3, 6 and 12 months
  MRI assessment of the volume
Efficacy of rapamycin on clinical symptoms | At 3, 6 and 12 months
  Clinical and fiberscopy evaluation by scoring
Pediatric Quality of Life Inventory (PedsQL 4) Scales | Baseline, at 3, 6 and 12 months
  Assesses health-related quality of life among children with chronic and acute diseases
Biological response to rapamycin | Baseline and at 6 months
  biological effect of mTOR blockage by measuring pAKT, p70S6 kinase, pMEK, and VEGF C, VEGFR3
Rapamycin side effects | Monthly during 1 years
  Side effect assessment using the NCI-CTC 3.0 scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fayoux, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hôpital Jeanne de Flandres, CHU, Lille
  - Hu Robert Debre Aphp - Paris, Paris

IPD SHARING:
Plan to Share IPD: No